CLINICAL TRIAL: NCT01122004
Title: The Effect of Gabapentin (Neurentin) and Pregabalin (Lyrica) in Pain Reduction After Photorefractive Keratectomy
Acronym: PRK
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shahid Beheshti University of Medical Sciences (Other)
Purpose: Treatment
Other Study IDs: 8877
Record Dates: First submitted 2010-04-12; First posted 2010-05-12 (Estimated); Last update posted 2010-05-12 (Estimated); Status verified 2010-03

CONDITIONS: Refractive Errors
MeSH Terms: conditions — Refractive Errors | interventions — Pregabalin

ARMS (2):
- Gabapentin (Active Comparator)
  Interventions: Drug: Pregabalin
- Pregabalin (Active Comparator)
  Interventions: Drug: Pregabalin

INTERVENTIONS:
Drug: Pregabalin
  Arms: Gabapentin
Drug: Pregabalin
  Arms: Pregabalin

SUMMARY:
The studied patients will be given randomly one of three following drugs1:Gabapentin2: Pregabalin or placebo for 3 days after Photorefractive keratectomy surgery. The pain will be measured based on visual analog scale(VAS) on the day of operation and on the 3 rd day (morning, evening) and then compared among three groups.

ELIGIBILITY:
Inclusion Criteria:

* patients candidate for PRK, 17<age<70

Exclusion Criteria:

* use of any systemic analgesic drugs, drug intolerance, need of systemic or topical administration of NSAIDs or eye drops for allergy and glaucoma, dry eyes, pregnancy, breast feeding

Min Age: 17 Years | Sex: All
Age Groups: Child, Adult, Older Adult

PRIMARY OUTCOMES:
pain degree based on visual analog scale(VAS)

CONTACTS AND LOCATIONS:
Locations (1):
- Ophthalmic Research Center, Tehran, Tehran Province, Iran